CLINICAL TRIAL: NCT05307510
Title: Influence of Custom Orthosis Post Carpometacarpal CMC) Arthroplasty
Brief Title: Influence of Custom Orthosis Post Carpometacarpal (CMC) Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UToledo301275
Record Dates: First submitted 2022-03-01; First posted 2022-04-01 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Thumb Osteoarthritis
Keywords: Carpometacarpal; Thumb; Arthroplasty; Splints; Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention A - prefabricated splint (Active Comparator): A prefabricated splint is provided to the client
  Interventions: Device: Prefabricated splint
- Intervention B - custom orthosis (Experimental): a custom orthosis (wrist splint with thumb spica) is fabricated by an occupational therapist
  Interventions: Device: Custom Orthosis

INTERVENTIONS:
Device: Prefabricated splint — Subjects will be provided either a prefabricated splint
  Arms: Intervention A - prefabricated splint
Device: Custom Orthosis — Subjects will be evaluated by an occupational therapist who will fabricate a custom orthosis.
  Arms: Intervention B - custom orthosis

SUMMARY:
This study aims to compare post-surgical outcomes of individuals who receive either a custom orthosis or prefabricated splint after carpometacarpal arthroplasty.

DETAILED DESCRIPTION:
This research study will randomly assign subjects post CMC arthroplasty to Intervention A (prefabricated splint) or Intervention B (custom orthosis). The orthosis and splint being used in this study are both considered standard practice. Subjects will be provided the splint or orthosis at the first post-operative appointment. Subjects who are assigned to Intervention A will be provided a pre-fabricated splint by a member of the surgical team. Subjects who are assigned to Invention B will be evaluated by an occupational therapist and a custom orthosis will be fabricated. Outcome measures include: QuickDASH, Pain Visual Analogue Scale, active range of motion measurements, the Applied Dexterity portion of the Arthritis Hand Function Test except for the putty cutting task, edema, Sandy Grading Score and the Orthotics and Prosthetics User's Survey (OPUS) Satisfaction with Device and Services. Data will be collected at the first, second, and third post-operative appointment.

ELIGIBILITY:
Inclusion Criteria:

* status post CMC arthroplasty
* 18 or older
* able to read and understand English
* capable of independently consenting to health care procedures.

Exclusion Criteria:

* if the surgeon identifies risk factors that would preclude random assignment to the control or experimental group
* if subject requests a prefabricated or custom orthosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Schmelzer, PhD, Principal Investigator — The University of Toledo
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for participants began in April of 2022 and concluded in September of 2023.
Period: Overall Study
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Started | 9 | 12
Data Collection I | 9 | 12
Data Collection II | 7 | 8
Data Collection III | 6 | 5
Completed | 6 | 5
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.78 (7.68) | 61.42 (8.93) | 62.86 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 7 | 11 | 18
  African American | 2 | 1 | 3
Sandy Grading Scale [Count of Participants; unit: Participants] — Description of wound dehiscence. Scale contains 6 grades (I, Ia, II, IIa, III, IIIa). I indicates no clinical signs of microbiological confirmation or infection.
  Participants
    Grade I | 9 | 12 | 21
    other grades | 0 | 0 | 0
VAS Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Pain Visual Analog Scale (VAS) is a self-report measure with a range of 0 = no pain to 10 = worst pain. Participants report pain at rest, in use, and at night.
  units on a scale
    Pain at rest | 4.11 (2.93) | 4.17 (2.76) | 4.14 (2.72)
    Pain at night | 4.89 (3.88) | 5.42 (2.94) | 5.19 (3.25)
    Pain in use | 7.67 (2.4) | 5.75 (1.82) | 6.57 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Post-operatively Using the Visual Analog Scale (Pain VAS)
Description: The Pain Visual Analog Scale is a self-report measure of pain with a range of 0= no pain - 10 = worst pain. Subjects report pain while using hand.
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
score on a scale
  Pain at rest | 2.5 (2.1) | 4.2 (1.3)
  Pain at night | 5.3 (.816) | 5.8 (2.6)
  Pain in use | 5 (2.76) | 6 (1.9)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Pain at rest; Test type: Superiority — Statistical analysis is under powered. N is too low; p = 0.135, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 2: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Pain at Night; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .716, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 3: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Pain in use; Test type: Superiority — Statistical Analysis underpowered. N is too small; p = .509, t-test, 2 sided — The threshold for statistical significance was p < 0.6

2. Primary Outcome: Change in Wound Dehiscence Post-operatively as Measured by Sandy Grading System
Description: Sandy Grading System is a scale used to measure wound dehiscence. Scale contains 6 grades (I, Ia, II, Ia, III, IIIa). A grade of I indicates no clinical signs of microbiological confirmation of infection and IIIa indicates presence of clinical signs and confirmed microbiological confirmation of infection. The higher number indicates increased presence of infection.
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
score on a scale | 1 (0) | 1 (0)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Test type: Superiority; p = 1, t-test, 2 sided

3. Secondary Outcome: Change in the Amount of Thumb CMC Active Range of Motion Post-operatively
Description: Goniometric measurements for active radial and palmar abduction will determine the amount of active movement. More range indicates better movement (0-50 = radial abduction norms) (0-70 = palmar abduction norms)
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
degrees
  Palmar Abduction | 37.50 (11.5) | 41 (12)
  Radial Abduction | 39.5 (7.1) | 42.6 (8.3)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Palmar abduction of surgical hand; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .635, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 2: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Radial Abduction Surgical Hand; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .521, t-test, 2 sided; Mean Difference (Net) = -3.1, 95% CI 2-sided [-13.6 to 7.4]

4. Secondary Outcome: Change in Client's Self-report of Hand Function Post-operatively as Measured by the QuickDash Disabilities of Arm, Shoulder, and Hand (QuickDASH)
Description: The QuickDash is a questionnaire about symptoms and ability to perform certain activities. Scores range from 0 (no disability) to 100 (severe disability).
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
score on a scale | 48 (15.6) | 40.6 (8.5)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .495, t-test, 2 sided; Mean Difference (Net) = 7.42, 95% CI 2-sided [-16.16 to 32.0]

5. Secondary Outcome: Change in the Degree of Dexterity Post-operatively as Measured by the Applied Dexterity Portion of the Arthritis Hand Function Test
Description: Four of Five items (fasten and unfasten buttons, lace a shoe and tie a bow, pin and unpin two safety pins in a cloth, pick up and manipulate four coins into a slot) will be completed. Each task will be timed. A shorter amount of time indicates better dexterity.
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
minutes
  Buttoning Buttons | .36 (.12) | .36 (.11)
  Lacing and tying a shoe | 1.37 (.22) | 1.35 (.35)
  Opening and closing safety pins | .31 (.13) | .33 (.05)
  Managing coins | .18 (.05) | .14 (.02)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Buttoning Buttons; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .953, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 2: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Lacing and tying a shoe; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .947, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 3: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Opening and closing safety pins; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .828, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 4: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Managing coins; Test type: Superiority — Statistical analysis is underpowered. N is too low; p = .169, t-test, 2 sided — The threshold for statistical significance was p < 0.6

6. Other Pre Specified Outcome: Patient Satisfaction With Device and Services as Measured by Orthotics and Prosthetics User's Survey (OPUS) Satisfaction With Device and Services
Description: A 21 item self-report questionnaire to measure satisfaction with device and services. Items 1-15 address services, items 16- 21 address device. Items are scored 0-4, with a higher score indicating higher satisfaction. Total score can range between 0-84.
Time Frame: 11-12 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 6 | 5
score on a scale
  Satisfaction with orthosis | 42.6 (9.85) | 45 (6.57)
  Satisfaction with services | 42 (4.76) | 45 (5.76)
Statistical Analysis 1: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Test type: Superiority — Statistical analysis underpowered. N too small; p = .917, t-test, 2 sided — The threshold for statistical significance was p < 0.6
Statistical Analysis 2: Comparison: Intervention A - Prefabricated Splint vs Intervention B - Custom Orthosis; Test type: Superiority — Statistical analysis is underpowered. N is too small; p = .837, t-test, 2 sided — The threshold for statistical significance was p < 0.6

7. Other Pre Specified Outcome: Change in Presence of Edema Post-operatively as Measured by a Circumferential Measurement
Description: A circumferential measurement at the base (metacarpal phalangeal joint) of the surgical thumb.
Time Frame: baseline (~10days after surgery), 5-6 week after surgery, 11-12 weeks after surgery
Population: Insufficient data to report. Circumferential measurement at base of thumb did not capture distal edema. Consequently, surgical team did not collect this data.
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: on average 12 weeks
Arm/Group | Intervention A - Prefabricated Splint | Intervention B - Custom Orthosis
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

LIMITATIONS AND CAVEATS:
The collaborating surgeon's standard practice patterns included the provision of a hand-based thumb orthosis at DC II. This unanticipated standard practice pattern significantly limits conclusions that can be drawn from the data regarding between group differences in the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT05307510/Prot_SAP_000.pdf